CLINICAL TRIAL: NCT06265389
Title: Pentoxifylline as an Adjuvant Therapy in the Treatment of Pediatric Pneumonia; A New Perspective of an Old Drug
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Rehab Zaki Elmeazawy, Doctor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pentoxifylline in pneumonia
Record Dates: First submitted 2024-02-11; First posted 2024-02-20 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Pentoxifylline as an Adjunct Therapy in the Treatment of Pneumonia
MeSH Terms: interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 50 children with community-acquired pneumonia will receive oral pentoxifylline in tablet form (Experimental): 50 children with community-acquired pneumonia will receive oral pentoxifylline in tablet form at a dose of 20 mg/kg/day, as an adjunct therapy to the usual pneumonia treatment for 5 days
  Interventions: Drug: Pentoxifylline Oral Tablet
- 50 children with community-acquired pneumonia with the standard pneumonia treatment. (No Intervention): 50 children with community-acquired pneumonia with the standard pneumonia treatment as a control group

INTERVENTIONS:
Drug: Pentoxifylline Oral Tablet — 50 children with community-acquired pneumonia will receive oral pentoxifylline in tablet form as an adjunct therapy to the usual pneumonia treatment for 5 days and the control group includes 50 children with community-acquired pneumonia with the standard pneumonia treatment.
  Other Names: TRENtal
  Arms: 50 children with community-acquired pneumonia will receive oral pentoxifylline in tablet form

SUMMARY:
Pentoxifylline is a xanthine-derived, commercially produced drug approved for the management of intermittent claudication in patients suffering from a chronic occlusive arterial disease of the limbs. Pentoxifylline has been documented to display anti-inflammatory and immunomodulatory effects, as well as some antithrombotic and antiviral effects. This drug has also been shown to reduce lung fibrosis in patients with COVID-19, as well as to prevent thromboembolic events. This work aims to assess the benefit of oral Pentoxifyllin supplementation, in addition to standard antibiotic and other supportive therapy, in the management of hospitalized children with community-acquired pneumonia

DETAILED DESCRIPTION:
This is a randomized clinical trial study that will be carried out on 100 children with Community-acquired pneumonia admitted to the Pulmonology Unit, Pediatric department.

Group 1: Pentoxifylline group, and group 2: Control group

ELIGIBILITY:
Inclusion Criteria:

* All children aged 2 months -18 years with community-acquired pneumonia diagnosed by signs and symptoms of CAP including; chest pain, dyspnea, tachypnea, or abnormal auscultatory findings plus focal findings on chest x-ray indicating community-acquired pneumonia

Exclusion Criteria:

* Children with immunodeficiency, chronic lung disease, malignancy, congenital lung anomalies, underlying disorders impacting respiration i.e. genetic, metabolic, neuromuscular disorders, and children with CHD affecting the pulmonary blood flow.

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Respiratory distress | 3 days
  Duration of improvement of respiratory distress
Temperature | 3 days
  Duration of defeverness
Oxygen saturation | 3 days
  Duration of normalization of hypoxia
CRP | 5 days
  Duration of normalization of CRP
LDH | 5 days
  Duration of normalization of LDH
D-dimer | 5 days
  Duration of normalization of D-dimer
Interleukin 6 | 5 days
  Duration of normalization of IL-6

SECONDARY OUTCOMES:
Hospital stays | 14 days
  Duration of stay in hospital
Pneumonia complications | 14 days
  Occurrence of pneumonia complications

OTHER OUTCOMES:
Surgical intervention | 14 days
  Intercostal chest tube, bronchoscope, decortication, lobectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No